CLINICAL TRIAL: NCT00405197
Title: Study on the Effect of Mono-Unsaturated Fatty Acids (MUFA) and the Mediterranean Diet on Hyperinsulinemia and Other Components of the Metabolic Syndrome
Brief Title: MARIS Study; Mediterranean Approach to Reduce Insulin-Resistance Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wageningen University (Other)
Collaborators: Netherlands Heart Foundation (Other); Unilever R&D (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: NHS 2003B068
Record Dates: First submitted 2006-11-28; First posted 2006-11-29 (Estimated); Last update posted 2007-12-12 (Estimated); Status verified 2007-12

CONDITIONS: Insulin Resistance; Metabolic Syndrome X; Dyslipidemia; Hypertension; Overweight
Keywords: MUFA; Mediterranean diet; Insulin resistance; metabolic syndrome X
MeSH Terms: conditions — Insulin Resistance; Metabolic Syndrome; Dyslipidemias; Hypertension; Overweight | interventions — Fatty Acids, Monounsaturated; Diet, Mediterranean

INTERVENTIONS:
Behavioral: Isocaloric diet high in MUFA or Mediterranean diet

SUMMARY:
Background: During the 1990s, the prevalence of the metabolic syndrome in the Netherlands ranged from 3% in women of 20-39 yrs to at least 33% in men 55 yrs and older and it is expected to increasing. Prevention is therefore warranted. In this respect the amount and type of fat in the diet deserves attention. Recently, an intervention study reported that a diet high in mono-unsaturated fatty acids (MUFA) such as from olive oil, increased insulin sensitivity in healthy subjects. However, additional beneficial effects can be expected from the Mediterranean diet as a whole. Hypothesis: Replacing saturated fatty acids (SFA) by mono-unsaturated fatty acids (MUFA) will improve hyperinsulinemia and dyslipidemia, and a typical Mediterranean diet will even have more pronounced effects. Study objectives: To investigate the impact of the Mediterranean diet, and especially the intake of MUFA, on markers of the metabolic syndrome in high-risk subjects. Methods: The controlled dietary intervention will include 60 subjects aged 40-65 years with moderate abdominal obesity. After a run-in diet for 2 weeks they will be assigned randomly to receive one of the three diets for a period of 8 weeks. Measurements of serum insulin concentration and other parameters will be carried out at weeks 2 and 10. Expected results: Our study will provide information on the role of MUFA and the expected beneficial impact of other factors of the Mediterranean type of diet on the metabolic syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Waist circumference ≥ 94 cm for men or ≥ 80 cm for women
* Age from 40 to 65 years at the time of randomisation
* Written informed consent obtained

Exclusion Criteria:

* Unable or unwilling to comply with study procedures.
* The use of drugs for lowering serum cholesterol, serum triglycerides, blood pressure, or diabetes.
* Unusual dietary patterns, including high alcohol intakes
* Recent (< 4 weeks) or current participation in a study with any investigational drug or dietary intervention.
* High concentrations of total cholesterol (>8 mmol/L).
* Diabetes mellitus.
* Being pregnant or giving breastfeeding.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2006-11; Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Fasting Insulin

SECONDARY OUTCOMES:
Systolic/ diastolic blood pressure
plasma glucose
serum HDL-cholesterol
serum triglycerides
waist-hip circumference
serum total cholesterol
serum LDL-cholesterol
Blood sample will be stored for measuring markers of inflammation.
Additionally in half of the subjects insulin sensitivity will be measured by the euglycemic hyperinsulinemic clamp.
Molecular markers in fat and muscle biopsies

CONTACTS AND LOCATIONS:
Overall Officials: Edith JM Feskens, Dr., Principal Investigator — Division of Human Nutrition, Wageningen University; Jeanne HM de Vries, Dr., Principal Investigator — Division of Human Nutrition, Wageningen University; Lisette CP de Groot, Prof., Principal Investigator — Division of Human Nutrition, Wageningen University; Lydia A. Afman, Dr., Principal Investigator — Division of Human Nutrition, Wageningen University; Michael R. Muller, Prof., Principal Investigator — Division of Human Nutrition, Wageningen University
Locations (2):
- Netherlands (2):
  - Hospital Gelderse Vallei, Ede
  - Wageningen University, Division of Human Nutrition, Wageningen

REFERENCES:
- [Background] Esposito K, Marfella R, Ciotola M, Di Palo C, Giugliano F, Giugliano G, D'Armiento M, D'Andrea F, Giugliano D. Effect of a mediterranean-style diet on endothelial dysfunction and markers of vascular inflammation in the metabolic syndrome: a randomized trial. JAMA. 2004 Sep 22;292(12):1440-6. doi: 10.1001/jama.292.12.1440. PMID 15383514
- [Background] Vessby B, Uusitupa M, Hermansen K, Riccardi G, Rivellese AA, Tapsell LC, Nalsen C, Berglund L, Louheranta A, Rasmussen BM, Calvert GD, Maffetone A, Pedersen E, Gustafsson IB, Storlien LH; KANWU Study. Substituting dietary saturated for monounsaturated fat impairs insulin sensitivity in healthy men and women: The KANWU Study. Diabetologia. 2001 Mar;44(3):312-9. doi: 10.1007/s001250051620. PMID 11317662
- [Background] Panagiotakos DB, Polychronopoulos E. The role of Mediterranean diet in the epidemiology of metabolic syndrome; converting epidemiology to clinical practice. Lipids Health Dis. 2005 Apr 12;4:7. doi: 10.1186/1476-511X-4-7. PMID 15826300
- [Background] Serra-Majem L, Roman B, Estruch R. Scientific evidence of interventions using the Mediterranean diet: a systematic review. Nutr Rev. 2006 Feb;64(2 Pt 2):S27-47. doi: 10.1111/j.1753-4887.2006.tb00232.x. PMID 16532897
- [Derived] van Dijk SJ, Feskens EJ, Bos MB, de Groot LC, de Vries JH, Muller M, Afman LA. Consumption of a high monounsaturated fat diet reduces oxidative phosphorylation gene expression in peripheral blood mononuclear cells of abdominally overweight men and women. J Nutr. 2012 Jul;142(7):1219-25. doi: 10.3945/jn.111.155283. Epub 2012 May 23. PMID 22623392
- [Derived] van Dijk SJ, Feskens EJ, Bos MB, Hoelen DW, Heijligenberg R, Bromhaar MG, de Groot LC, de Vries JH, Muller M, Afman LA. A saturated fatty acid-rich diet induces an obesity-linked proinflammatory gene expression profile in adipose tissue of subjects at risk of metabolic syndrome. Am J Clin Nutr. 2009 Dec;90(6):1656-64. doi: 10.3945/ajcn.2009.27792. Epub 2009 Oct 14. PMID 19828712